CLINICAL TRIAL: NCT04851067
Title: Dry Needling Versus Manual Therapy in Patients With Mechanical Neck Pain: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hendricks Regional Health (Other)
Responsible Party: Principal Investigator, Jeevan Pandya, PT,MHS, OCS, COMT, FAAOMPT, Hendricks Regional Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-10
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling and Therapeutic Exercises (DNTEx) (Active Comparator): Dry Needling - A fine needle, of 5-10 mm, will be used to penetrate the skin, subcutaneous tissues, and muscle with the intent to stimulate Myofascial Trigger Point (MTrP) or mechanically disrupt tissue without the use of an anesthetic.
  Therapeutic Exercises - Are exercises will be performed to achieve a specific physical benefit, including increasing and maintaining range of motion, strengthening weak muscles, increasing joint flexibility, or improving cardiovascular and respiratory function.
  Interventions: Other: Dry Needling and Therapeutic Exercises (DNTEx)
- Manual Therapy and Therapeutic Exercises (MTTEx) (Active Comparator): Joint Mobilization - A manual therapy technique comprising of a continuum of skilled passive movements to the joint complex will be applied at varying speeds and amplitudes. It will include a low-grades/velocity (grades I and II), high grades (grades III and IV), and small- or large-amplitude passive movement techniques within the patient's physiological range of motion and within the patient's control with the intent to restore optimal motion, function, and/ or to reduce pain.
  Joint Manipulation - A passive, high velocity, low amplitude thrust will be applied to a localized joint segment/s within its anatomical limit with the intent to restore optimal motion, function, and/ or to reduce pain.
  Interventions: Other: Manual Therapy and Therapeutic Exercises (MTTEx)

INTERVENTIONS:
Other: Dry Needling and Therapeutic Exercises (DNTEx) — Already included in arm/group descriptions.
  Arms: Dry Needling and Therapeutic Exercises (DNTEx)
Other: Manual Therapy and Therapeutic Exercises (MTTEx) — Already included in arm/group descriptions.
  Arms: Manual Therapy and Therapeutic Exercises (MTTEx)

SUMMARY:
Background: The current physical therapy evidence for treating patients with the mechanical neck pain recommends both, manual therapy (MT) and dry needling (DN) along with cervical and scapulothoracic exercises.1 However, at present, investigators still don't have any evidence suggesting if one treatment approach, the manual therapy and exercises or dry needling and exercises, is superior to the other in treating patients with the mechanical neck pain. Objective: The aim of this study is to compare the effects of dry needling and manual therapy on pain, disability, range of motion, strength, and patient perceived improvements in the patients with mechanical neck pain. Methods: Investigators will conduct a randomized, single-blind, placebo-controlled trial in accordance with the CONSORT guidelines. Patients with primary complain of neck pain, with a minimum score of 2 on Numeric Pain Rating Scale (NPRS), a minimum of 10 points or 20% score of Neck Disability Index (NDI), and who are over the age of 18 will be enrolled in the study. Subjects with any red flags, history of surgery at the cervical or thoracic spine, neurological symptoms, nerve root compression, whiplash in the last 6 weeks, pending legal actions related to neck pain, on workers compensation, insufficient English language skills, and/or contraindications to dry needling or manual therapy, will be excluded from the study. A total of 75 patients will be recruited for the study, who will be randomized to two groups - (1) Dry Needling and Therapeutic Exercises (DNTEx) and (2) Manual Therapy and Therapeutic Exercises (MTTEx). All participants will be treated for seven physical therapy treatment sessions of 30 minutes each over a maximum of 6 weeks. The primary outcome measure will NDI, which will evaluate disability of patients. While secondary outcome measures would be: NPRS (score range from 0 to 10) to assess pain, Patient-Specific Functional Scale [PSFS], (score ranges from 3 to 30) will measure a patient-specific measure of function important significant to them, Range of Motion (ROM) will measure changes in the motion of flexion, extension, bilateral rotation, and bilateral side-bending at the cervical spine, The Neck Flexor Endurance Test (NFET) will measure the improvement in the endurance of neck flexor muscles, Fear Avoidance Belief Questionnaire (FABQ) will measure patients' fear of pain with movements and resulting avoidance of physical activity because of their fear, and The Patient Global Rating of Change (GROC) will measure each patient's self-perceived improvement. An assessor, who is blinded to the group allocation, will collect all outcome measures at baseline, 2weeks, discharge session/7th treatment session, and 3 months after discharge/7th treatment session. An a priori alpha level of 0.05 will be used for all analyses. Investigators will examine the primary aim with a repeated-measures analysis of covariance (ANCOVA), using pretest scores as covariates, with treatment groups (Dry needling + Exercise Vs. MT + Exercise) as the between subjects' independent variables and time (baseline, 2 weeks, Discharge [7 sessions], 12 weeks post discharge) as the within-subjects independent variable. The hypothesis of interest is the 2-way group * time interaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Primary complaint of neck pain
3. Neck Disability Index > 10 points=20%

Exclusion Criteria:

1. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e., tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, symptoms of vertebrobasilar insufficiency, pregnancy, cervical spinal stenosis, bilateral upper extremity symptoms etc.
2. Use of blood thinners
3. History of whiplash injury within the past six weeks
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e., positive Hoffman's and/or Babinski reflexes), etc.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   1. Muscle weakness involving a major muscle group of the upper extremity
   2. Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps)
   3. Diminished or absent sensation to pinprick in any upper extremity dermatome
6. Prior surgery to the neck or thoracic spine
7. Workers' compensation or pending legal action regarding their neck pain
8. Insufficient English language skills to complete all questionnaires
9. Inability to comply with treatment and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 0 Week
  The NDI is used to measure pain-related disability associated with activities of daily living in people with neck pain. The NDI contains 10 items-7 related to activities of daily living, 2 related to pain, and 1 related to concentration. Each item is scored on a 6-point scale, from 0 to 5; therefore, the maximum score is 50. The total score is expressed as a percentage (total possible score, 100%), with higher scores corresponding to greater disability.9,77 Content, construct validity, and reliability of the NDI has been previously shown in patients with neck pain. The NDI has been used by researchers to evaluate the effect of treatments on patients' perceived levels of functioning and disability. The NDI has showed good reliability and validity in patients with mechanical neck pain.
Neck Disability Index | 2 Weeks
  The NDI is used to measure pain-related disability associated with activities of daily living in people with neck pain. The NDI contains 10 items-7 related to activities of daily living, 2 related to pain, and 1 related to concentration. Each item is scored on a 6-point scale, from 0 to 5; therefore, the maximum score is 50. The total score is expressed as a percentage (total possible score, 100%), with higher scores corresponding to greater disability.9,77 Content, construct validity, and reliability of the NDI has been previously shown in patients with neck pain. The NDI has been used by researchers to evaluate the effect of treatments on patients' perceived levels of functioning and disability. The NDI has showed good reliability and validity in patients with mechanical neck pain.
Neck Disability Index | 4 Weeks
  The NDI is used to measure pain-related disability associated with activities of daily living in people with neck pain. The NDI contains 10 items-7 related to activities of daily living, 2 related to pain, and 1 related to concentration. Each item is scored on a 6-point scale, from 0 to 5; therefore, the maximum score is 50. The total score is expressed as a percentage (total possible score, 100%), with higher scores corresponding to greater disability.9,77 Content, construct validity, and reliability of the NDI has been previously shown in patients with neck pain. The NDI has been used by researchers to evaluate the effect of treatments on patients' perceived levels of functioning and disability. The NDI has showed good reliability and validity in patients with mechanical neck pain.
Neck Disability Index | 12 Weeks post discharge
  The NDI is used to measure pain-related disability associated with activities of daily living in people with neck pain. The NDI contains 10 items-7 related to activities of daily living, 2 related to pain, and 1 related to concentration. Each item is scored on a 6-point scale, from 0 to 5; therefore, the maximum score is 50. The total score is expressed as a percentage (total possible score, 100%), with higher scores corresponding to greater disability.9,77 Content, construct validity, and reliability of the NDI has been previously shown in patients with neck pain. The NDI has been used by researchers to evaluate the effect of treatments on patients' perceived levels of functioning and disability. The NDI has showed good reliability and validity in patients with mechanical neck pain.

SECONDARY OUTCOMES:
Numeric pain Rating Scale (NPRS) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  The number that the respondent indicates on the scale to rate their pain intensity is recorded. Scores range from 0-10. In a 11-point numeric scale, 0 represents "NO PAIN" and 10 represents "EXTREME PAIN" (e.g., "pain as bad as you can imagine" and "worst pain imaginable"). The NPRS has been shown to be reliable and valid.
Patient Specific Functional Scale (PSFS) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  The PSFS focuses on the patient's opinion of their function and requires the physiotherapist to ask the patient to list three activities that are limited by the condition for which they are seeking treatment, the overall PSFS score is an average of all three activities scores. Patients select a value that best describes their current activity level on a 11-point scale. On this 11-point scale (0 represents - "unable to perform" and 10 represents - "able to perform at prior level").
Global Rating of Change Scale (GROC) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  It is used to measure each patient's self-perceived improvement.87 The GROC will be used, which is a 15-point global rating scale described by Jaeschke et al.87 The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). The global rating will be administered at the follow-up examinations only.
Cervical Range of Motion (CROM) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  Cervical Range of motion is the extent of movement of the joints in the cervical spine, which measured in degrees.88,89 Movements are measured in flexion, extension, rotation, and side bending by an inclinometer and goniometer.88 Normal CROM are - 60-80 degree of flexion, 60 degree of extension, 45 degree side bending, and 90 degree of rotation.
Fear Avoidance Belief Questionnaire (FABQ) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  It measure patients' fear of pain with movements and resulting avoidance of physical activity because of their fear.90, 91 The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two sub-scales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24).
The Neck Flexor Endurance Test (NFET) | 0 week, 2 weeks, 4 weeks, and 12 weeks post discharge
  It assess the endurance in the endurance of neck flexor muscles.92 The test is performed with a patient in a supine, hook-lying position. Patient maximally retracts the chin and holds it isometrically. Then, patient lifts the head and neck 1-inch (2.5cm) off the table, while keeping the chin retracted to the chest. The therapist places a hand on the table just below the occipital bone of the patient's head and focuses on the skin folds along the patient's neck. Therapist can give verbal commands (such as - "Tuck your chin", "Hold your head up", "keep your chin tucked", etc.), when either the skin fold(s) begins to separate, or the patient's occiput touches the therapist's hand. The test is terminated if the skin fold(s) is separated due to loss of chin tuck or the patient's head touches the therapist's hand for more than 1 second. Normal Values are - Men: 38.9 seconds, Women: 29.4 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cleland, PT, PHD, Study Chair — Tuft's University; Shane Koppenhaver, PT, PHD, Study Director — Robbins College of Health and Human Sciences, Baylor University; Louie Puentedura, PT, PHD, Study Director — Robbins College of Health and Human Sciences, Baylor University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pandya J, Puentedura EJ, Koppenhaver S, Cleland J. Dry Needling Versus Manual Therapy for Patients With Mechanical Neck Pain: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2024 Apr;54(4):267-278. doi: 10.2519/jospt.2024.12091. PMID 38284367